CLINICAL TRIAL: NCT02868840
Title: Evaluating the Effect of Tai Chi Applied Stroke Rehabilitation on Physical and Cognitive Functioning
Brief Title: Tai Chi for Stroke Rehabilitation on Balance and Cognition
Acronym: TCSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Rhayun Song, Professor, Chungnam National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChungnamNU
Record Dates: First submitted 2016-07-27; First posted 2016-08-16 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Stroke
Keywords: stroke; Tai ji; postural balance; cognition
MeSH Terms: conditions — Stroke | interventions — Aquatic Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi group (Experimental): Tai Chi exercise, twice a week, one hour per session. participated in Tai Chi either while seated or standing upon their comfort level.
  Interventions: Behavioral: Tai Chi exercise
- Symptom management group (Active Comparator): manage stroke symptom through phone and text message along with other rehabilitation therapy.
  Interventions: Behavioral: symptom management

INTERVENTIONS:
Behavioral: Tai Chi exercise — exercise twice a week each for one hour
  Other Names: seated Tai Chi
  Arms: Tai Chi group
Behavioral: symptom management — sending text message weekly to manage symptoms related to stroke
  Other Names: message counselling
  Arms: Symptom management group

SUMMARY:
Tai Chi, an ancient Chinese martial art, is a low intense aerobic exercise characterized by continuous movements that embrace the mind, body, and spirit. Tai Chi addresses the integration and balance of mind and body using the fundamental principles of slow, smooth, and continuous movement control, and the transfer of body weight while maintaining an upright and relaxed posture. The present randomized clinical trial project aims to apply the suggested principles as the typical features of Tai Chi applied stroke rehabilitation, and to evaluate the effects on physical (balance), psychological, and cognitive function.

DETAILED DESCRIPTION:
Cerebrovascular disease is a major global concern. The individuals with stroke would suffer from disease associated symptoms which influence their functioning in everyday life. These symptom clusters were usually known to be sharing similar underlying mechanisms. It is clear that the development of effective stroke rehabilitation involves interdisciplinary team approach to manage physical, social, cognitive, and psychological functioning in this population.

Tai Chi, an ancient Chinese martial art, is a low intense aerobic exercise characterized by continuous movements that embrace the mind, body, and spirit. Tai Chi addresses the integration and balance of mind and body using the fundamental principles of slow, smooth, and continuous movement control, and the transfer of body weight while maintaining an upright and relaxed posture. The newly developed style of Tai Chi for health programs is the seated Tai Chi, which shares the common Tai Chi principles while being modified to adjust the movements for patients with limited mobility.

The present randomized clinical trial project aims to apply the suggested principles as the typical features of Tai Chi applied stroke rehabilitation, and to evaluate the effects on physical (balance), psychological, and cognitive function. Only a few studies ever addressed the feasibility of Tai Chi for stroke rehabilitation, and the relationship between cognition and balance in this population is still very early stage of investigation. The main purpose of our collaborating project is to explore the direct relationship between cognition and balance in stroke patients during their rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as stroke at least for 3 months upto 2 years
* eligible to participate rehabilitation therapy referred by primary physician

Exclusion Criteria:

* not able to understand questionnaires
* not able to stand alone for balance test

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
balance | 3 months, 6 months
  postural stability test will be measured by standard computerized test

SECONDARY OUTCOMES:
activities of daily living | 3 months, 6 months
  activities of daily living will be measured by Modified rankin scale
knee muscle strength | 3 months, 6 months
  knee flexor and extensor strength by isokinetic testing measured by Biodex

OTHER OUTCOMES:
cognition | 3 months, 6 months
  measured by Korean version of Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Rhayun Song, PhD, Principal Investigator — Chungnam National University
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen BL, Guo JB, Liu MS, Li X, Zou J, Chen X, Zhang LL, Yue YS, Wang XQ. Effect of Traditional Chinese Exercise on Gait and Balance for Stroke: A Systematic Review and Meta-Analysis. PLoS One. 2015 Aug 20;10(8):e0135932. doi: 10.1371/journal.pone.0135932. eCollection 2015. PMID 26291978
- [Background] Tao J, Rao T, Lin L, Liu W, Wu Z, Zheng G, Su Y, Huang J, Lin Z, Wu J, Fang Y, Chen L. Evaluation of Tai Chi Yunshou exercises on community-based stroke patients with balance dysfunction: a study protocol of a cluster randomized controlled trial. BMC Complement Altern Med. 2015 Feb 25;15:31. doi: 10.1186/s12906-015-0555-1. PMID 25888114